CLINICAL TRIAL: NCT02799758
Title: Efficacy & Long-term Safety Comparison Study of NK-104-CR & Livalo® IR With Primary Hyperlipidemia or Mixed Dyslipidemia
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Kowa Research Institute, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NK-104-CR-3.02US
Record Dates: First submitted 2016-06-10; First posted 2016-06-15 (Estimated); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Hyperlipidemia; Dyslipidemia
MeSH Terms: conditions — Hyperlipidemias; Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NK-104-CR (Experimental): NK-104-CR 8 mg tablet and Placebo (for Livalo® IR 4 mg tablet) orally once daily for 52 weeks.
  Interventions: Drug: NK-104-CR; Drug: Placebo (for Livalo® IR)
- Livalo® IR (Active Comparator): Livalo® IR 4 mg tablet and Placebo (for NK-104-CR 8 mg tablet) orally once daily for 52 weeks.
  Interventions: Drug: Livalo® IR; Drug: Placebo (for NK-104-CR)

INTERVENTIONS:
Drug: NK-104-CR — NK-104-CR 8 mg for 52 weeks
  Arms: NK-104-CR
Drug: Livalo® IR — Livalo® IR 4 mg daily for 52 weeks
  Arms: Livalo® IR
Drug: Placebo (for NK-104-CR) — NK-104-CR 8 mg placebo for 52 weeks
  Arms: Livalo® IR
Drug: Placebo (for Livalo® IR) — Livalo® IR 4 mg placebo for 52 weeks
  Arms: NK-104-CR

SUMMARY:
The purpose of this study is to demonstrate the superior efficacy of NK-104-CR 8 mg daily compared to Livalo® IR 4 mg daily on fasting serum low-density lipoprotein cholesterol (LDL-C) reduction and to evaluate the comparative safety of NK-104-CR 8 mg daily to Livalo® IR 4 mg daily after long-term treatment

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with primary hyperlipidemia or mixed dyslipidemia
* Patients for whom lipid-lowering therapy is indicated according to NCEP ATPIII
* Patients who are naïve to statin or who are able to safely discontinue the use of all lipid-lowering agents for 4 weeks before randomization and throughout study participation

Exclusion Criteria:

* Homozygous familial hypercholesterolemia;
* Any conditions which may cause secondary dyslipidemia.
* Newly diagnosed or poorly controlled diabetes mellitus as defined by HbA1c >9%

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-02; Primary Completion 2017-07 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Percent change in Low-density lipoprotein cholesterol (LDL-C) | Baseline to Week 12 endpoint

CONTACTS AND LOCATIONS:
Locations (69):
- United States (69):
  - Foley, Alabama
  - Huntsville, Alabama
  - Montgomery, Alabama
  - Muscle Shoals, Alabama
  - Little Rock, Arkansas
  - Greenbrae, California
  - Huntington Park, California
  - Lomita, California
  - Long Beach, California
  - Los Angeles, California
  - Santa Ana, California
  - Spring Valley, California
  - Tustin, California
  - Walnut Creek, California
  - Milford, Connecticut
  - Atlantis, Florida
  - Cooper City, Florida
  - Coral Springs, Florida
  - Fleming Island, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Oviedo, Florida
  - Dawsonville, Georgia
  - Macon, Georgia
  - Suwanee, Georgia
  - Addison, Illinois
  - Chicago, Illinois
  - Gurnee, Illinois
  - Morton, Illinois
  - Evansville, Indiana
  - Topeka, Kansas
  - Louisville, Kentucky
  - Owensboro, Kentucky
  - Oxon Hill, Maryland
  - Biloxi, Mississippi
  - Olive Branch, Mississippi
  - Jefferson City, Missouri
  - St Louis, Missouri
  - Omaha, Nebraska
  - Manlius, New York
  - High Point, North Carolina
  - Salisbury, North Carolina
  - Wilmington, North Carolina
  - Winston-Salem, North Carolina
  - Fargo, North Dakota
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Franklin, Ohio
  - Oklahoma City, Oklahoma
  - Medford, Oregon
  - Beaver, Pennsylvania
  - Harleysville, Pennsylvania
  - Jersey Shore, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Moncks Corner, South Carolina
  - Simpsonville, South Carolina
  - Summerville, South Carolina
  - Austin, Texas
  - Houston, Texas
  - Katy, Texas
  - Plano, Texas
  - Round Rock, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Richmond, Virginia
  - Suffolk, Virginia
  - Seattle, Washington
  - Kenosha, Wisconsin